CLINICAL TRIAL: NCT07264504
Title: Experimentation of Formaldehyde Purification by Plants in the Anatomy and Cytology Department
Acronym: DETOXANAPATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0095
Record Dates: First submitted 2025-05-06; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Formaldehyde; Pathological Anatomy and Cytology
Keywords: formaldehyde; plants; pathological anatomy and cytology; remediation; purification; occupational exposure; occupational health; carcinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laboratory staff (Experimental): Before / after installation of plants
  Interventions: Biological: Biological measurement of urinary formic acid; Other: Plant installation

INTERVENTIONS:
Biological: Biological measurement of urinary formic acid — Biological measurement of urinary formic acid
Other: Plant installation — plant installation

SUMMARY:
Formaldehyde is notably used as a tissue fixator in pathological anatomy. Despite its toxicity, it continues to be widely used because it is currently not substitutable. Some plants have shown their ability to absorb formaldehyde. The investigators would like to show if the installation of plants in the Anatomy and Cytology Department of the Amiens University Hospital reduces the exposure to formaldehyde of the staff of this department. After carrying out atmospheric and biological measurements the investigators will install 15 plants in both rooms where the staff is most exposed to formaldehyde : the macroscopy room and the reception room. The atmospheric and biological measurements will be redone after two months.

ELIGIBILITY:
Inclusion Criteria:

* To work in the Department of Pathological Anatomy and Cytology
* Adult (> 18 years old)
* Patient information and collection of non-opposition

Exclusion Criteria:

* Pregnant woman
* Patients under guardianship or safeguarding of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Atmospheric formaldehyde concentration | 2 months
  Variation of Atmospheric measurement of formaldehyde between before and after plant installation

SECONDARY OUTCOMES:
Variation of urinary formic acid concentration | 2 months
  Variation of Biological measurement of urinary formic acid between before and after plant installation

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No